CLINICAL TRIAL: NCT04095650
Title: A New Model to Reach Vulnerable Older Adults With Pain Self-management Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH); American Pain Society (Other)
Responsible Party: Principal Investigator, Mary Janevic, Assistant Research Scientist, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00154949; K01AG050706 (NIH)
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will engage in a 7-week chronic pain self-management program.
  Interventions: Behavioral: STEPS (Seniors using Technology to Engage in Pain Self-management)

INTERVENTIONS:
Behavioral: STEPS (Seniors using Technology to Engage in Pain Self-management) — Participants will meet with a community health worker (CHW) at a one-hour in-person study orientation session. At this session, they will be introduced to the program, learn how to use the online modules and associated materials, and schedule six weekly telephone sessions with the CHW. Participants will be given a wearable physical activity tracker to use throughout the course of the program. They can choose to report daily step counts by automatically syncing to an app or via text message. Each week during the study period, participants will engage with content on the website, have a session with the community health worker, track their daily steps, and set and work toward pain-management goals.

SUMMARY:
Learning chronic pain self-management skills can help patients improve daily functioning and quality of life, while avoiding risks associated with opioids and other pharmacological treatments. Community health workers (CHWs) may help make chronic pain self-management interventions more accessible to older adults living in underserved communities. The goal of this study is to conduct a feasibility test of a chronic pain self-management intervention delivered by CHWs, in conjunction with mobile health tools, in a sample of 25 older adults recruited from community sites in Detroit, Michigan. This study will involve the use of mixed quantitative and qualitative methods to assess participant engagement and satisfaction, and change in pain-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English-proficient
* Age >= 60 years
* Ambulatory with or without assistive device
* Community-living
* Have a cell or landline phone
* Have Internet access (home or elsewhere)
* Self-reported chronic musculoskeletal pain (pain in muscles or joints for > 3 months); >4 (0-10 scale) average pain level over last week; >1 day/previous 30 when pain made it difficult to do usual activities
* Ability to attend a one-time study orientation session

Exclusion Criteria:

* Serious acute illness or hospitalization in last month
* Planned surgery in next three months
* Significant cognitive impairment as indicated by affirmative response to question: "Do you have significant difficulties with your memory that get in the way of your usual daily activities?"
* Other severe physical or psychiatric disorder judged by study team to pose significant barrier to deriving program benefit.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Change in pain interference | baseline and 8 weeks
  The Pain Interference 6-item subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS)-43 Adult Profile. Items ask how much pain in the last 7 days has interfered with daily activities such as household chores and social activities (1=not at all to 5=very much); raw total scale scores range from 6 (low interference) to 30 (high interference)..
Participant engagement | 8 weeks
  Number of completed sessions with the community health worker (range 1 to 7).

SECONDARY OUTCOMES:
Participant Global Impression of Change | 8 weeks
  Two items: 1) How participant thinks their pain has changed from baseline (much worse (-3) to much better(+3)). 2) How participant thinks their functioning has changed from baseline (much worse (-3) to much better(+3)).
Participant satisfaction: Likert-scale questions | 8 weeks
  Likert-scale questions about participant satisfaction with the program; e.g., whether participation increased understanding of pain management (Strongly Agree=1 to Strongly Disagree=5), and with selected program elements (e.g., community health workers, videos, website).

CONTACTS AND LOCATIONS:
Overall Officials: Mary Janevic, PhD, Principal Investigator — University of Michigan School of Public Health
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT04095650/ICF_000.pdf